CLINICAL TRIAL: NCT02151773
Title: Freeze-dried Live Attenuated Measles and Rubella Combined Vaccine "Takeda" Special Drug Use Surveillance of Vaccinees After the First Vaccination
Brief Title: Freeze-dried Live Attenuated Measles/Rubella Combined Vaccine (Schwarz FF-8 Strain/TO-336 Strain) Special Drug Use Surveillance of Vaccinees After the First Vaccination
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: 247-011; JapicCTI-142490 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Measles/Rubella
Keywords: Pharmacological therapy
MeSH Terms: conditions — Measles; Rubella

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Live attenuated measles/rubella combined vaccine: Live attenuated measles/rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) is dissolved in 0.7 milliliter (mL) of accompanying reconstitution fluid (water for injection [Japanese Pharmacopoeia]), and a 0.5-mL portion is typically administered subcutaneously as a single dose.
  Interventions: Drug: Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain)

INTERVENTIONS:
Drug: Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) — Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain)
  Other Names: Freeze-dried live attenuated measles and rubella combined vaccine "Takeda"

SUMMARY:
The purpose of this survey is to assess the safety freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) (freeze-dried live attenuated measles and rubella combined vaccine "Takeda") in terms of the occurrence of unknown/known adverse drug reactions and factors that may influence the safety of vaccinees after the first vaccination.

DETAILED DESCRIPTION:
This survey was designed to assess the safety of live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) (freeze-dried live attenuated measles and rubella combined vaccine "Takeda") in terms of the occurrence of unknown/known adverse drug reactions and factors that may influence the safety of vaccinees after the first vaccination.

Freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) is dissolved in 0.7 mL of accompanying reconstitution fluid (water for injection [Japanese Pharmacopoeia]), wherein a 0.5-mL portion is typically administered subcutaneously as a single dose.

In addition, freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) should be used in accordance with the "Regulations for Vaccination" and the "Guidelines for Routine Vaccination."

ELIGIBILITY:
Inclusion Criteria:

-Vaccinees who meet both of the following conditions [1] and [2]:

1. Vaccinees who have no prior history of either measles or rubella vaccination and who received freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) as the initial vaccination.
2. Vaccinees whose guardians are able to participate in a questionnaire survey on the health status of vaccinees after vaccination with freeze-dried live attenuated measles and rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain).

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Measles/rubella
Sampling Method: Non-Probability Sample
Enrollment: 3493 (Actual)
Dates: Start 2006-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Postmarketing Group Manager, Study Chair — Takeda

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 152 investigative sites in Japan from 07 February 2006 to 30 April 2009.
Pre-assignment Details: Participants with a historical diagnosis of measles/rubella who received live attenuated measles/rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) as per routine medical practice were observed in this study.
Groups:
- Live Attenuated Measles/Rubella Combined Vaccine: Participants receiving freeze-dried live attenuated measles/rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) 0.5 milliliter (mL), injection, subcutaneously as a single dose as per routine medical practice were observed.
Period: Overall Study
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Started | 3493
Completed | 3429
Not Completed | 64
Not completed — Protocol Deviation | 64

BASELINE CHARACTERISTICS:
Population: Analysis set included all participants who were enrolled and completed the study.
Groups:
- Live Attenuated Measles/Rubella Combined Vaccine: Participants receiving freeze-dried live attenuated measles/rubella combined vaccine (Schwarz FF-8 strain/TO-336 strain) 0.5 mL, injection, subcutaneously as a single dose as per routine medical practice were observed.
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Number analyzed (Participants) | 3429
Age, Customized [Number; unit: participants]
  >=12 to less than (<)18 months | 2921
  Greater than or equal to (>=) 18 months | 508
Gender [Count of Participants; unit: Participants]
  Female | 1670
  Male | 1759
Region of Enrollment [Number; unit: participants]
  Japan | 3429
Predisposition to hypersensitivity [Number; unit: participants] — Participants may be represented in more than 1 category.
  participants
    Drug hypersensitivity | 10
    Food hypersensitivity | 187
    Other hypersensitivity | 23
    Not determined | 41
Complications [Number; unit: participants] — Complications defined as a disease or a health condition for each participant at the start of study. Complications were classified as congenital anomalies, endocrine disorders, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, gastrointestinal (GI) disorders, renal disease and other complications. Other complications included all complications except for those mentioned above. Participants may be represented in more than 1 category.
  participants
    Congenital anomalies | 20
    Endocrine disorders | 1
    Hematologic disorders | 8
    Psychiatric and nervous system disorders | 18
    Cardiovascular disorders | 14
    Respiratory disorders | 139
    GI disorders | 11
    Renal disease | 4
    Other complications | 120
Medical history [Number; unit: participants] — Medical history defined as a disease or a health condition for each participant before start of the study. Medical history was classified as congenital anomalies, hematologic disorders, psychiatric and nervous system disorders, cardiovascular disorders, respiratory disorders, GI disorders, hepatic and biliary disorders, renal disease and other medical history. Other medical history included all medical history except for those mentioned above. Participants may be represented in more than 1 category.
  participants
    Congenital anomalies | 19
    Hematologic disorders | 10
    Psychiatric and nervous system disorders | 54
    Cardiovascular disorders | 25
    Respiratory disorders | 149
    GI disorders | 49
    Hepatic and biliary disorders | 3
    Renal disease | 2
    Other medical history | 177
Concomitant medication [Number; unit: participants] — Participants may be represented in more than 1 category.
  participants
    Not determined or not described | 10
    Antibiotic drugs | 17
    Neuropsychiatric drugs | 5
    GI drugs | 21
    Other concomitant medication | 117
Items that require careful examination before vaccination [Number; unit: participants] — Participants were analyzed for any underlying disease such as cardiovascular disease. Allergy related to the components of the freeze-dried live attenuated measles and rubella combined vaccine was reported. Participants may be represented in more than 1 category.
  participants
    Underlying disease | 48
    Pyrexia and generalized rash | 4
    History of convulsions | 33
    Allergy to components of study vaccine | 49
Experience with other vaccine [Number; unit: participants]
  Prior exposure to vaccine | 3315
  No prior exposure to vaccine | 92
  Not determined or not described | 22
Type of surveying method after vaccination [Number; unit: participants] — Type of surveying method after vaccination included questionnaire, consultation and other survey (for example, call). Participants may be represented in more than 1 category.
  participants
    Questionnaire | 3149
    Consultation | 1230
    Other survey | 154

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Serious Adverse Drug Reactions
Description: Serious adverse drug reactions are defined as serious adverse events (SAE) which are in the investigator's opinion of causal relationship to the study treatment. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Frequency of adverse events and factors that may influence safety were not to be assessed as endpoints of this study and were registered as endpoints by mistake. Instead, adverse drug reactions were assessed as endpoint.
Time Frame: Baseline up to Day 28
Population: Safety analysis set included all participants who received at least one dose of study vaccination.
Measure: Number; unit: participants
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Number analyzed (Participants) | 3369
participants | 7

2. Secondary Outcome: Number of Participants Reporting One or More Adverse Drug Reactions
Description: Adverse drug reactions are defined as adverse events (AE) which are in the investigator's opinion of causal relationship to the study treatment. AE are defined as any unfavorable and unintended signs, symptoms or diseases temporally associated with the use of a medicinal product reported from the first dose of study drug to the last dose of study drug.
Time Frame: Baseline up to Day 28
Population: Safety analysis set included all participants who received at least one dose of study vaccination.
Measure: Number; unit: participants
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Number analyzed (Participants) | 3369
participants | 1183

ADVERSE EVENTS:
Time Frame: Baseline up to Day 28
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. Only adverse drug reactions were collected in this study.
Arm/Group | Live Attenuated Measles/Rubella Combined Vaccine
Serious Adverse Events (participants affected / at risk) | 7/3369
Other Adverse Events (participants affected / at risk) | 1181/3369
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Live Attenuated Measles/Rubella Combined Vaccine (N=3369)
Exanthema subitum (Infections and infestations) | 1
Convulsion (Nervous system disorders) | 3
Kawasaki's disease (Vascular disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 2
Pyrexia (General disorders) | 5
White blood cell count increased (Investigations) | 1
C-reactive protein increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Live Attenuated Measles/Rubella Combined Vaccine (N=3369)
Mood altered (Psychiatric disorders) | 132
Cough (Respiratory, thoracic and mediastinal disorders) | 307
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 436
Diarrhoea (Gastrointestinal disorders) | 178
Rash (Skin and subcutaneous tissue disorders) | 316
Injection site erythema (General disorders) | 141
Pyrexia (General disorders) | 633

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.